CLINICAL TRIAL: NCT04728360
Title: A Multicenter, Randomized, Double-Blind, Parallel-Arm, Phase 3 Study to Compare Efficacy and Safety of BAT2206 With Stelara® in Patients With Moderate to Severe Plaque Psoriasis
Brief Title: Comparative Study of BAT2206 With Stelara® in Patients With Moderate to Severe Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bio-Thera Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BAT-2206-002-CR
Record Dates: First submitted 2021-01-24; First posted 2021-01-28 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2022-08

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BAT2206 (Experimental): Patients who weigh ≤ 100 kg: BAT2206 45 mg (1 injection of 45 mg/0.5 mL) by SC injection via PFS.
  Patients who weigh > 100 kg: EU-sourced Stelara 90 mg (2 injections of 45 mg/0.5 mL each) by SC injection via PFS.
  Interventions: Drug: BAT2206
- Stelara (EU-sourced) (Active Comparator): Patients who weigh ≤ 100 kg: EU-sourced Stelara 45 mg (1 injection of 45 mg/0.5 mL) by SC injection via PFS.
  Patients who weigh > 100 kg: EU-sourced Stelara 90 mg (2 injections of 45 mg/0.5 mL each) by SC injection via PFS.
  Interventions: Drug: Stelara (EU-sourced)

INTERVENTIONS:
Drug: BAT2206 — 45 mg/0.5 mL
  Arms: BAT2206
Drug: Stelara (EU-sourced) — 45 mg/0.5 mL
  Arms: Stelara (EU-sourced)

SUMMARY:
This study is a multicenter, randomized, double-blind, parallel-arm, Phase 3 study designed to compare efficacy, safety, immunogenicity, and PK of BAT2206 with Stelara in patients with moderate to severe plaque psoriasis.

The study is composed of a ≤ 28-day screening period, a 16-week initial treatment period (TP1), a 24-week secondary treatment period (TP2), a 12-week efficacy and safety follow-up period up to end-of-study visit, for a maximum total study duration of 56 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years old with a diagnosis of plaque-type psoriasis for at least 24 weeks before screening.
2. Have moderate to severe plaque-type psoriasis as defined at screening and baseline by:

   1. PASI ≥ 12,
   2. sPGA ≥ 3, and
   3. body surface area affected by chronic plaque-type psoriasis ≥ 10%
3. Failed to respond to, or have a contraindication to, or is intolerant to other systemic therapies including cyclosporine, methotrexate or psoralen and ultraviolet (UV) A
4. Female patients of childbearing potential and male patients with a female partner of childbearing potential must be willing to use a highly effective contraceptive precaution throughout the study period and continuing for at least 15 weeks after the last dose of study drug. See APPENDIX 1 for the acceptable highly effective contraceptive methods. Abstinence from heterosexual intercourse is accepted when this is the usual lifestyle of the patient and must be continued for at least 15 weeks after the last dose of study drug. A female patient is considered not of childbearing potential when postmenopausal (at least 12 consecutive months without menses without an alternative medical cause) or surgically sterilized (hysterectomy, bilateral salpingectomy, and bilateral oophorectomy).
5. If female of childbearing potential, patient should have a negative pregnancy test result at screening and baseline visits.
6. Must be willing to provide written consent and to comply with the requirements of the study protocol.

Exclusion Criteria:

1. Have any forms of psoriasis at the time of the screening visit other than plaque-type such as erythrodermic psoriasis, pustular psoriasis, guttate psoriasis, medication-induced psoriasis or other skin conditions (eg, eczema) that would interfere with evaluations of the effect of investigational product on psoriasis.
2. Have previously received ustekinumab, a biosimilar of ustekinumab, or any drug that targets interleukin-12 or interleukin-23.
3. Have received any biologic agents other than those prohibited (see exclusion #2) within 12 weeks or 5 half-lives (whichever is longer) before the baseline visit.
4. Have received topical therapies for the treatment of psoriasis (such as corticosteroids, vitamin D analogs, or retinoids) within 2 weeks before baseline visit.
5. Have received UVA phototherapy (with or without oral psoralen), UVB phototherapy, any systemic steroids or nonbiological drugs for the treatment of psoriasis within 4 weeks before baseline visit
6. Have received any investigational drug within 8 weeks or 5 half-lives (whichever is longer) before baseline visit
7. Have received any herbal remedies or traditional medicines used to treat psoriasis within 4 weeks before baseline visit
8. History of allergy to the active substance or any of the excipients of study drugs, or of hypersensitivity to latex.
9. History of invasive infection (eg, histoplasmosis, coccidioidomycosis, blastomycosis).
10. Presence of active infection at screening, history of infection requiring intravenous antibiotics and/or hospitalization ≤ 8 weeks before baseline visit or oral antibiotics ≤ 2 weeks before baseline visit. Minor fungal infections may be allowed.
11. Any recurrent bacterial, fungal, or viral infection that, (based on the investigator´s clinical assessment), makes the patient unsuitable for the study, including recurrent/disseminated herpes zoster.
12. Meet any of the following criteria relative to latent or active tuberculosis (TB) infection.
13. Evidence of malignancy, lung infection, or abnormalities suggestive of active TB on chest radiography (x-ray or computed tomography) performed within 12 weeks before the screening visit or during the screening period.
14. Any history of malignancy or lymphoproliferative disease at any time, except curative treatment for nonmelanoma skin cancer or resected carcinoma in situ of the cervix.
15. Have a transplanted organ/tissue or stem cell transplantation.
16. Have an underlying metabolic, hematologic, renal, hepatic, pulmonary, neurologic, endocrine, cardiac, infectious, or gastrointestinal condition, which in the opinion of the investigator places the patient at unacceptable risk.
17. Have a history of demyelinating diseases (including myelitis) or neurologic symptoms suggestive of demyelinating disease.
18. Any major surgical procedure within 12 weeks of the baseline visit or planned during the study.
19. History of clinically significant drug or alcohol abuse in the last 12 months as judged by the investigator.
20. Pregnant or breastfeeding (lactating) women.
21. Patient is considered by the investigator, for any reason, to be an unsuitable candidate for the study.
22. Patients participating in another investigational drug or device (a device is an instrument, apparatus, implement, machine, contrivance, or implant, including a component part or accessory intended for use in the diagnosis of disease or other conditions, or in the cure, mitigation, treatment, or prevention of disease) trial or planning on participating in another clinical trial during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 556 (Actual)
Dates: Start 2021-07-06 (Actual); Primary Completion 2022-10-12 (Actual); Study Completion 2023-07-07 (Actual)

PRIMARY OUTCOMES:
PASI | 0-12 weeks
  Percent improvement from baseline in Psoriasis Area and Severity Index (PASI) score to Week 12

SECONDARY OUTCOMES:
PASI score | Weeks 4, 8, 16, 20, 28, 40, and 52
  Percent improvement from baseline in PASI score to Weeks 4, 8, 16, 20, 28, 40, and 52
PASI-50/75/90/100 | Weeks 4, 8, 12, 16, 20, 28, 40, and 52
  Proportion of patients who achieve at least 50/75/90/100% improvement from baseline in PASI (PASI-50/75/90/100) at Weeks 4, 8, 12, 16, 20, 28, 40, and 52
Static Physician's Global Assessment (sPGA) score | Weeks 4, 8, 12, 16, 20, 28, 40, and 52
  Change from baseline in static Physician's Global Assessment (sPGA) score to Weeks 4, 8, 12, 16, 20, 28, 40, and 52

CONTACTS AND LOCATIONS:
Overall Officials: Min Zheng, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided